CLINICAL TRIAL: NCT07285447
Title: Re-use of Ambu aScope During Exploration of the Common Bile Duct for Stones in Low-Resource Settings- a Retrospective Study
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Abhijeet Kumar, Associate Professor, B.P. Koirala Institute of Health Sciences
Other Study IDs: IRC/2994/025
Record Dates: First submitted 2025-09-26; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: CBD Stone
Keywords: Ambu aScope; Choledochoscope; CBD (Common Bile Duct) exploration; Laparoscopic; Open; Low-resource settings
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- use of Ambu aScope during open and laparoscopic CBD exploration
  Interventions: Device: Ambu aScope for visualization of biliary tree during exploration of CBD for stone

INTERVENTIONS:
Device: Ambu aScope for visualization of biliary tree during exploration of CBD for stone — Ambu aScope, in stead of choledochoscope in low-reource settings, can be used for visualization of biliary tree and retrieval of stone during surgical open or laparoscopic exploration of CBD

SUMMARY:
Various methods confirm stone clearance during surgical exploration of bile duct, but choledochoscopy is considered the most effective. However, choledochoscopes are expensive and often unavailable in low-resource settings. The Ambu aScope, a disposable flexible video-bronchoscope used in anesthesia, has been successfully tried as a cheaper alternative for CBD (Common Bile Duct) exploration in other countries. In Nepal, where affordability is a concern, reuse of properly disinfected Ambu aScopes may be justifiable if proven safe. Existing studies are limited and small in scale; this study is the first from Nepal to evaluate the reuse of Ambu aScope for choledochoscopy.

This retrospective observational study will include all patients with CBD stones who underwent CBD exploration for stone using Ambu aScope in Department of Surgery of BPKIHS, Dharan between January 2022 and December 2024.

Case record files of all patients who underwent CBD exploration using aScope as a Choledochoscope over last 3 years period will be obtained from medical record section and computer database of our department. All relevant information including patient demographics, indication for a CBD exploration, operative approach and procedure performed, intraoperative achievement of acceptable view of extrahepatic biliary tree using an aScope, intraoperative stone clearance on direct visualization of biliary tree and confirmation on postoperative T-tube cholangiogram or imaging on 10-14th postoperative day and intra/post-operative complications associated with the use of the aScope will be entered in a preformed proforma. In case of some missing information in medical case report sheet or computer database of our department, patient will be called directly on the contact number provided in admission sheet and through the telephonic conversation, the concerned queries will be cleared. Data will be entered in Microsoft Excel and analyzed by SPSS version 29.0.1.0. Qualitative data were described using numbers and percentages. Quantitative data will be described using range (minimum and maximum), mean, standard deviation, and median.

ELIGIBILITY:
Inclusion Criteria:

* all patients with CBD stones who underwent CBD exploration for stone using the Ambu aScope in Department of Surgery of BPKIHS, Dharan between January 2022 and December 2024

Exclusion Criteria:

* Single stone of <1cm, Patient not fit for general anesthesia, Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with CBD stones who underwent CBD exploration for stone using the Ambu aScope in Department of Surgery of BPKIHS, Dharan between January 2022 and December 2024
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2025-08-13 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of re-use of aScope during exploration of CBD for stone | intraoperative and early post operative upto 2 weeks
  Success rate (in percentage) of achieving acceptable view of extrahepatic biliary tree form the 2nd generation biliary radicles proximally to the ampulla of Vater distally with Ambu aScope.
  Stone clearance rate (in percentage) with the use of ambu aScope
  Occurrence (in terms of percentage) of complications (such as Injury to biliary tree, Cholangitis related with reuse of the aScope)

SECONDARY OUTCOMES:
Demographic distribution of patients with CBD stone | perioperative period upto 2weeks post-surgery
  Demographic distribution (in terms of mean age, gender, and stone characteristics) of patients who underwent CBD exploration using aScope as a choledochoscope

CONTACTS AND LOCATIONS:
Locations (1):
- B. P. Koirala Institute of Health Science, Dharān, Province No-1, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chuang KT, Chuang SC, Kuo KK, Chang WT, Chuang SH, et al. (2024) Laparoscopic vs. Open Choledocholithiasis Interventions: Unraveling the Dominant Trends in Surgical Practice: A Single-Center, 6-Year, Retrospective Study. J Surg 9: 11089 https://doi.org/10.29011/2575-9760.
- [Result] Yi HJ, Hong G, Min SK, Lee HK. Long-term Outcome of Primary Closure After Laparoscopic Common Bile Duct Exploration Combined With Choledochoscopy. Surg Laparosc Endosc Percutan Tech. 2015 Jun;25(3):250-3. doi: 10.1097/SLE.0000000000000151. PMID 25856136
- [Result] Daniel C, Pereira J, Prudente C, Constantino J, Sa M, Casimiro C. Laparoscopic choledochoscopy with Ambu(R) aScope 3 in the treatment of coledocholithiasis: a series of cases. J Surg Case Rep. 2018 Mar 29;2018(3):rjy046. doi: 10.1093/jscr/rjy046. eCollection 2018 Mar. PMID 29977501
- [Result] Aawsaj YM, Ibrahim IK, Gilliam A. Novel method for laparoscopic common bile duct exploration performed using a disposable bronchoscope (Ambu® aScope TM). Kurdistan J Appl Res. 2017; 2: 49-51.
- [Result] Samir M, Selima M, Hefzy M. Choledochoscopy using disposable bronchoscope Ambu aScope 3: a single-institute experience. The Egyptian Journal of Surgery. 2022; 40(3). doi: 10.4103/ejs.ejs_166_21